CLINICAL TRIAL: NCT05563883
Title: Atrial Fibrillation and Cancer: a Nationwide French Cohort Study
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Caen (Other)
Collaborators: University Hospital, Tours (Other)
Responsible Party: Principal Investigator, Joachim ALEXANDRE, Prof, University Hospital, Caen
Other Study IDs: PMSI_092022
Record Dates: First submitted 2022-09-24; First posted 2022-10-03 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Atrial Fibrillation; Cancer; Thromboembolism; Bleeding
MeSH Terms: conditions — Atrial Fibrillation; Neoplasms; Thromboembolism; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: event occurence — occurence of an event of interest: (AF, cancer, thromboembolism, bleeding, mortality...

SUMMARY:
Atrial fibrillation (AF) is a common complication associated with cancer but the risk of AF according to the cancer localization and status as well as the risk of thromboembolisms, bleedings and mortality are poorly known.

The objective of this study is to use a very large French nationwide cohort to adress thèses questions.

ELIGIBILITY:
Inclusion Criteria:

* adult hospitalized patients
* with an ICD-10 code discharge from january 2010 to december 2019 in the French national hospital discharge database (PMSI Programme de Médicalisation des Systèmes d'Information)

Exclusion Criteria:

* children

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized from january 2010 to december 2019 and having an available ICD-10 code discharge.
Sampling Method: Non-Probability Sample
Enrollment: 5000000 (Estimated)
Dates: Start 2022-09-22 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
atrial fibrillation | from inclusion in the cohort up to 10 years
  occurrence of atrial fibrillation
cancer | ffrom inclusion in the cohort up to 10 years
  occurrence of cancer

SECONDARY OUTCOMES:
thromboembolism | from inclusion in the cohort up to 10 years
  occurrence of thromboembolism
bleeding | from inclusion in the cohort up to 10 years
  occurrence of bleeding
mortality | from inclusion in the cohort up to 10 years
  occurrence of mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Cardiologie, Centre Hospitalier Universitaire Trousseau, Tours, France